CLINICAL TRIAL: NCT07366034
Title: A Study to Evaluate the Dose-exposure, Safety, and Exploratory Efficacy of Nerandomilast in Children and Adolescents From 2 Years to Less Than 18 Years of Age With Fibrosing Interstitial Lung Disease (Part A: Double-blind, Placebo-controlled in Children From 6 to Less Than 18 Years of Age and Open-label Active Treatment in Children From 2 to Less Than 6 Years of Age), Followed by an Open-label Phase With Active Treatment (Part B)
Brief Title: A Study to Find Out How Nerandomilast is Tolerated, Handled by the Body, and if it Helps Children and Adolescents With Interstitial Lung Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0022; 2025-523369-32-00 (Registry Identifier: CTIS); 1111-1326-6351 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2026-01-23; First posted 2026-01-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Fibrosing Interstitial Lung Disease

STUDY DESIGN:
Intervention Model Description: Part A:
  * double-blind, placebo-controlled in children from 6 to less than 18 years of age
  * and open-label active treatment in children from 2 to less than 6 years of age
  Part B:
  - open-label phase with active treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking applies to double-blind part of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants aged 2 to <6 years (Experimental): Part A and Part B: Nerandomilast (open-label)
  Interventions: Drug: Nerandomilast
- Participants aged 6 to <18 years, group 1 (Experimental): Part A: Nerandomilast (blinded), Part B: Nerandomilast (open-label)
  Interventions: Drug: Nerandomilast
- Participants aged 6 to <18 years, group 2 (Experimental): Part A: Placebo (blinded), Part B: Nerandomilast (open-label)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nerandomilast — Nerandomilast
  Other Names: JASCAYD®
  Arms: Participants aged 2 to <6 years; Participants aged 6 to <18 years, group 1
Drug: Placebo — Placebo
  Arms: Participants aged 6 to <18 years, group 2

SUMMARY:
This study is open to children and adolescents aged 2 to 17 years with interstitial lung disease (ILD). Nerandomilast has just been approved in some countries to help adults with a lung condition called idiopathic pulmonary fibrosis. The purpose of this study is to understand how nerandomilast is tolerated and handled by the body and whether nerandomilast also helps children and adolescents with ILD.

For participants aged 6 to 17 years when joining, the study has 2 parts. In the first part, participants are put into 1 of 2 groups randomly, which means by chance. One group gets nerandomilast and the other group placebo. Placebo looks like nerandomilast but does not contain any medicine.

Participants are twice as likely to be in the nerandomilast group. They take tablets twice a day for 6 months. After these 6 months, in the second part of this study, they get nerandomilast for at least 2 years regardless of what they got in the first part.

Young participants aged 2 to 5 years when joining get nerandomilast from the start. They receive tablets twice a day for at least 2 and a half years.

Depending on when a person joins, the study lasts between 2 and a half years and up to 5 years. During this time, participants may visit the study site about 18 to 30 times. Study doctors collect blood samples to check participants' health and to find out how their body handles the study medicine. Doctors also check the function of the lungs, body growth, and how participants feel. The study doctors also regularly check participants' health and take note of any changes. For participants aged 6 to 17 years, the results are compared between the groups to see whether nerandomilast treatment helps children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 2 to <18 years old at Visit 2.
* Participants with evidence of fibrosing ILD on high-resolution computed tomography (HRCT) within 12 months of Visit 1 as assessed by the investigator and confirmed by central review.
* For children ≥6 years: Participants with forced vital capacity (FVC) % predicted ≥25% at Visit 2.
* Participants with clinically significant fibrosing ILD at Visit 2, as assessed by the investigator based on any of the following:

  * Fan score ≥3, or
  * Documented evidence of clinical progression over time based on either

    * a 5-10% relative decline in FVC % predicted accompanied by worsening symptoms, or
    * a ≥10% relative decline in FVC % predicted, or
    * increased fibrosis on HRCT, or
    * other measures of clinical worsening attributed to progressive lung disease (e.g. increased oxygen requirement, decreased diffusion capacity).

Further inclusion criteria apply.

Exclusion Criteria:

* Previous treatment with nerandomilast.
* Participants treated with other oral/systemic PDE4 and non-selective PDE inhibitors within 30 days before Visit 1.
* Participants treated with pirfenidone in the 8 weeks prior to Visit 1.
* Unstable pulmonary arterial hypertension (PAH).
* Active vasculitis, unstable or uncontrolled within 8 weeks prior to Visit 1 or during the screening period.
* Any suicidal behaviour (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour) in the past (lifetime).
* Any suicidal ideation of type 4 or 5 on the columbia suicidal severity rating scale (C-SSRS) in the past 3 months at Visit 1 or at Visit 2 (i.e. active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, intent, and plan).
* Participants with clinically significant depression symptoms defined as the short version of mood and feeling questionnaire (SMFQ) score ≥8.

Further exclusion criteria apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2029-04-27 (Estimated); Study Completion 2031-04-14 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration curve (AUC) T,SS based on sampling at steady state using rich sampling in participants from 6 years to less than 18 years and sparse sampling in participants younger than 6 years | At week 2 in Part A and Week 28 in Part B
Occurrence of a treatment-emergent adverse event | up to Week 26

SECONDARY OUTCOMES:
Absolute change from baseline in oxygen saturation (SpO2) [%] on room air at rest | at Week 26 and Week 52
Absolute change from baseline in height [cm] | at Week 26 and Week 52
Absolute change from baseline in pediatric quality of life inventory (PedsQL™) | at Week 26 and Week 52
  Health-related quality of life will be assessed in children using the PedsQL™ questionnaire. For younger children who are unable to perform self-assessment, a parent proxy may be required. The score ranges from 0-100, a higher score indicates a better health related quality of life.
Occurrence of a treatment-emergent adverse event (Yes/No) over the whole trial | up to 5 years
Time to first respiratory-related hospitalisation [days] over the whole trial | up to 5 years
Time to first acute interstitial lung disease (ILD) exacerbation or death [days] over the whole trial | up to 5 years
Time to death [days] over the whole trial | up to 5 years
Participant acceptability based on number/size of tablets | at Week 2 and Week 26
  Acceptability is defined as the overall ability and willingness of the participant to use the medicinal product as intended.
  Assessment of acceptability will be performed by the participant using the acceptability questionnaire.
Participant acceptability based on the use of the dispenser | at Week 2 and Week 26
Absolute change from baseline in FVC [% predicted] (applicable to participants ≥6 years) | at Week 26 and Week 52
Absolute change from baseline in 6-min walk distance [m] (applicable to participants ≥6 years) | at Week 26 and Week 52

CONTACTS AND LOCATIONS:
Locations (41):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Argentina (2):
  - Fundacion Respirar, CABA
  - Hospital de Pediatria Prof. Dr. Juan P. Garrahan, CABA
- Brussels - UNIV HUDERF, Brussels, Belgium
- Brazil (4):
  - Serviços Medicos Respirar Sul Fluminense, Barra Mansa
  - Associação dos Funcionários Públicos do Estado do Rio Grande do Sul - Hospital Ernesto Dorneles, Porto Alegre
  - IMIP Pernambuco, Recife
  - Centro de Pesquisa Clinica do Instituto da Crianca - HCFMUSP, São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada
- China (3):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Hunan Provincial People's Hospital, Changsha
  - The Children's Hospital of Fudan University, Shanghai
- University Hospital Motol, Prague, Czechia
- Aarhus University Hospital, Aarhus N, Denmark
- Finland (2):
  - HUS Lasten ja nuorten sairaudet, Kliinisen tutkimuksen yksikkö, Helsinki
  - Tampere University Hospital, Tampere
- France (5):
  - HOP Femme Mère Enfant, Bron
  - HOP Intercommunal, Créteil
  - HOP Timone, Marseille
  - HOP Armand-Trousseau, Paris
  - HOP Necker - Enfants Malades, Paris
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Hamburger Zentrum für Kinder- und Jugendrheumatologie, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Aristotle University, Thessaloniki, Thessaloniki, Greece
- Italy (2):
  - Istituto G. Gaslini, Genova
  - Osp. Pediatrico Bambin Gesù, Roma
- Japan (2):
  - Osaka Women's and Children's Hospital, Osaka, Izumi
  - National Center for Child Health and Development, Tokyo, Setagaya-ku
- Centro de Investigacion Clinica y Medicina Traslacional (CIMeT), Guadalajara, Mexico
- Amsterdam University Medical Center, Amsterdam, Netherlands
- University Clinical Center of the Medical University of Warsaw, Warsaw, Poland
- ULS de Santa Maria, E.P.E, Lisbon, Portugal
- Spain (2):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency